CLINICAL TRIAL: NCT02433522
Title: Extended Follow Up of the Mainritsan 2 Study. Comparison Between a Long Term and a Conventional Maintenance Treatment With Rituximab: a Placebo- Controlled Randomized Trial
Brief Title: Comparison Between a Long Term and a Conventional Maintenance Treatment With Rituximab
Acronym: MAINRITSAN3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Roche Pharma AG (Industry); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P110146 extended; 2012-001963-66 (EudraCT Number)
Record Dates: First submitted 2015-03-23; First posted 2015-05-05 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: ANCA-associated Vasculitides
Keywords: ANCA-associated vasculitides; Maintenance treatment; Rituximab; Granulomatosis with polyangiitis; Microscopic polyangiitis
MeSH Terms: conditions — Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Granulomatosis with Polyangiitis; Microscopic Polyangiitis | interventions — Rituximab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rituximab (Experimental): 500 mg rituximab infusion at the randomization visit and every 6 months for 18 months
  Interventions: Drug: rituximab
- Placebo (Placebo Comparator): Placebo infusion at the randomization visit and every 6 months for 18 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: rituximab — 500 mg rituximab infusion at the randomization visit and every 6 months for 18 months. Each infusion will be preceded by an infusion of 1000 mg paracetamol, 100 mg methylprednisolone and 5 mg dexchlorpheniramine.
  Arms: Rituximab
Drug: Placebo
  Arms: Placebo

SUMMARY:
MAINRITSAN study compared Rituximab and azathioprine as maintenance therapy for ANCA-associated vasculitides. In this study, Rituximab (5 infusions at D1, D15, M6, M12, M18) was superior to azathioprine (2 mg/kg/day) to prevent relapses of AAV 28 months after the inclusion (Guillevin et al. NEJM 2014). Nevertheless, in the follow-up study of MAINRITSAN, up to 30% of patients experienced a relapse 38 months after the last rituximab infusion (unpublished data). Right now, no randomized controlled study has been carried in order to evaluate the best duration of the maintenance treatment with rituximab.

The investigators objective is to evaluate the efficacy of a long term rituximab treatment to prevent relapses of ANCA-associated vasculitis in patients in remission after a first phase of rituximab maintenance treatment.

The investigators will conduct a randomized placebo-controlled trial of a long term rituximab maintenance treatment (46 months) against a conventional maintenance treatment (18 months).

ELIGIBILITY:
Inclusion Criteria:

First, patients must have been included in MAINRITSAN 2 and in addition to meeting the criteria for inclusion and non-inclusion.

MAINRITSAN 2 inclusion criteria:

* Granulomatosis with Polyangiitis Or microscopic polyangiitis complying Or kidney-limited disease With or without detectable ANCA (anti-neutrophil cytoplasmic antibodies) at the time of diagnosis or relapse, and at remission.
* Who have achieved remission using a treatment combining corticosteroids and an immunosuppressive agent, including corticosteroids, cyclophosphamide IV or oral (the use of another immunosuppressant is allowed, according to the current French guidelines, as well as plasma exchanges and/or IV immunoglobulins, or rituximab).
* Interval of 1 month between the end of the immunosuppressant treatment and the randomization time if cyclophosphamide or methotrexate were used, interval between 4 and 6 months if rituximab was used
* Age > 18 years without age limit higher when the diagnosis is confirmed.
* Informed and having signed the consent form to take part in the study.

and Patients must meet all of the following criteria:

* In complete remission (BVAS 0) at 28 months of MAINRITSAN2 study.
* Informed patient who accepted to participate in MAINRITSAN 2 and who signed the informed consent to this extension.
* Randomized on the day of the evaluation of the primary endpoint of MAINRITSAN 2 during the visit M28 (last visit of the protocol).

Exclusion Criteria:

* Eosinophilic granulomatosis with polyangiitis (EGPA)
* History of severe allergic manifestations or anaphylactic manifestations following humanized or murine monoclonal antibodies infusions
* Pregnant or breast feeding women. Contraception is required for women who could be pregnant during treatment follow up and during the year following the last infusion.
* Infection by HIV (positive serology), HCV (positive serology), or HBV (HBsAg positive or anti-HBc antibody positive with anti-HBs antibody negative)
* Uncontrolled infection at time of inclusion in the extended follow-up study.
* Other severe bacterial, viral , mycobacterial or fungal infection(s), occurring within the last 3 months before of randomization. A severe infection is defined by the hospitalization, a life or organ threatening.
* Severe chronic obstructive bronchopathy (FEV < 50% or dyspnea stage III).
* Cardiac failure, stage IV according to the NYHA classification.
* Recent history of coronary artery disease (<1 month).
* Ongoing malignancy or hematologic disease within 5 years before inclusion.
* Patient with severe immunodepression characterized by clinical manifestations.
* Participation to another concomitant therapeutic study (except observational studies or studies without therapeutic intervention).
* Psychiatric disease that may interfere with the study.
* Non affiliation to a health insurance.
* Uncontrolled severe cardiac disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2015-03-31 (Actual); Primary Completion 2018-08-16 (Actual); Study Completion 2018-08-16 (Actual)

PRIMARY OUTCOMES:
Vasculitis score 2003 (BVAS 2003 ) | 28 months
  Relapse free survival rates (BVAS > 0)

SECONDARY OUTCOMES:
Number of adverse events, | 28 months
  adverse events including infectious effects and their severity in each arm
number of patients experiencing at least one adverse event in both arms | 28 months
correlation of ANCA level with the clinical events | 28 months
ANCA level during follow-up | 28 months
correlation B-Lymphocytes CD-19 level with the clinical events | 28 months
B-Lymphocytes CD-19 level during follow-up | 28 months
number of B memory cells during follow-up in both arms | 28 months
correlation number of B memory cells with the clinical events | 28 months
Number of patients with ANCA in each arm | 28 months
Time frame to death in both arms | 28 months
time frame of first minor relapse | 28 months
time frame of first major relapse | 28 months
  "the reappearance of disease activity or worsening, with a Birmingham Vasculitis Activity Score >0, and involvement of one or more major organs, disease-related life-threatening events, or both"
Cumulated dose of corticosteroid treatment | 28 months
Number and severity of damages | 28 months
number of of gammaglobulins | 28 months
Quality of life : SF36 (The Short Form (36) Health Survey) | 28 months
functional capacities : HAQ (Health Assessment Questionnaire ) | 28 months

CONTACTS AND LOCATIONS:
Overall Officials: Loic GUILLEVIN, MD-PhD, Study Chair — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hopital cochin, Paris, France

REFERENCES:
- [Background] Pagnoux C, Guillevin L; French Vasculitis Study Group; MAINRITSAN investigators. Rituximab or azathioprine maintenance in ANCA-associated vasculitis. N Engl J Med. 2015 Jan 22;372(4):386-7. doi: 10.1056/NEJMc1414728. No abstract available. PMID 25607433
- [Result] Charles P, Perrodeau E, Samson M, Bonnotte B, Neel A, Agard C, Huart A, Karras A, Lifermann F, Godmer P, Cohen P, Hanrotel-Saliou C, Martin-Silva N, Pugnet G, Maurier F, Sibilia J, Carron PL, Gobert P, Meaux-Ruault N, Le Gallou T, Vinzio S, Viallard JF, Hachulla E, Vinter C, Puechal X, Terrier B, Ravaud P, Mouthon L, Guillevin L; French Vasculitis Study Group. Long-Term Rituximab Use to Maintain Remission of Antineutrophil Cytoplasmic Antibody-Associated Vasculitis: A Randomized Trial. Ann Intern Med. 2020 Aug 4;173(3):179-187. doi: 10.7326/M19-3827. Epub 2020 Jun 2. PMID 32479166